CLINICAL TRIAL: NCT02679105
Title: Intralymphatic Immunotherapy in Increasing Doses up to 10 000 SQ-U -a Human Randomized Clinical Trial
Brief Title: Intralymphatic Immunotherapy in Increasing Doses, After Subcutaneous Immunotherapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other); Skane University Hospital (Other); Sodra Alvsborgs Hospital (Other)
Responsible Party: Principal Investigator, Lars Olaf Cardell, Professor, Head of Division, MD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-001259-63
Record Dates: First submitted 2016-01-23; First posted 2016-02-10 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Rhinitis, Allergic
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALK diluent (Placebo Comparator): Human albumin
  Interventions: Drug: ALK diluent
- ALK Alutard birch or 5-grasses (Active Comparator): Grass pollen suspension or birch pollen suspension
  Interventions: Drug: ALK Alutard birch or 5-grasses

INTERVENTIONS:
Drug: ALK Alutard birch or 5-grasses — 3 injections with 4-5 weeks interval.
  Other Names: ALK Alutard birch pollen or ALK Alutard grass pollen; ATC-code V01AA, V04CL and V07AB
  Arms: ALK Alutard birch or 5-grasses
Drug: ALK diluent — 0,3% human albumin
  Other Names: Human albumin
  Arms: ALK diluent

SUMMARY:
The study evaluates the safety and effect of intralymphatic allergen specific immunotherapy in increasing doses. Patients that have already undergone subcutaneous immunotherapy will be treated with three intralymphatic injections in increasing doses; 1000 SQ-U, 3000 SQ-U and 10 000 SQ-U, or placebo.

DETAILED DESCRIPTION:
38 patients with seasonal allergic rhinitis that have recently (within 20 months) ended a full subcutaneous immunotherapy protocol with birch or grass allergen with improvement but not full symptom relief are recruited. Study subjects are randomized to intralymphatic injections with placebo or ALK Alutard 5-grasses or birch.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55
* Accepted and signed informed consent.
* Recently (within 20 months) ended a full 3 year program with subcutaneous immunotherapy (SCIT) with amelioration of symptoms but not full symptom relief.

Exclusion Criteria:

* Previously subcutaneous immunotherapy (SCIT) with total symptom relief.
* Previously SCIT but no symptom improvement at all.
* Sensitizations to house dust mite or furry animals, with symptoms.
* Severe atopic dermatitis.
* Patients with significant diseases other than allergic rhinitis. A significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study.
* Patients with a respiratory tract infection in the past 4 weeks prior to Visit 2.
* Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception (i.e., oral contraceptives, intrauterine devices, diaphragm, or subdermal implants).
* Known autoimmune or collagen disease
* Cardiovascular disease
* Perennial pulmonary disease including asthma
* Hepatic disease
* Known renal insufficiency
* Cancer
* Hematologic disease
* Chronic infectious disease
* Any medication with a possible side-effect of interfering with the immune response
* Previous immuno- or chemotherapy, apart from SCIT
* Disease or conditions rendering the treatment of anaphylactic reactions difficult (symptomatic coronary heart diseases, severe arterial hypertension and treatment with β-blockers)
* Major metabolic disease
* Known or suspected allergy to the study product
* Obesity with BMI > 30 since subcutaneous fat makes ultrasound imaging of lymph nodes harder which may risk the correct placement of injection.
* Patients who, in the opinion of the investigator, abuse alcohol or drugs within 2 years prior to Visit 1.
* Patients who have taken an investigational drug within 1 month or six half lives, whichever is greater, prior to Visit 1.
* Mental incapability of coping with the study
* Withdrawal of informed consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2015-05; Primary Completion 2016-10 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Total daily symptoms and medications score | 5-7 months after treatment
  Difference between active and placebo group in total daily symptoms and medications score during the pollen season.

SECONDARY OUTCOMES:
Improvement on Visual Analogue Scale (VAS) | During pollen season and recalled after pollen season, approximately 1 year after the start of treatment.
  Difference in improvement on VAS between active and placebo group.
Change in skin prick test reactivity | 4-8 weeks after treatment, 9-12 months after treatment
  Tested with ALK Soluprick. Measured as the wheal area in millimeter for birch- or grass pollen.
Change in symptoms score after nasal allergen challenge | 4-8 weeks after treatment, 9-12 months after treatment
  0,1 ml of ALK Aquagen Birch or Timothy 10 000 SQU/ml is deposited in each nostril and allergy symptoms are recorded.
Difference between active and placebo group in Quality of Life measured with Juniper Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) | Up to 7 months after treatment.
  At peak pollen season after treatment.
Difference between active and placebo group in Quality of Life measured with Sino Nasal Outcome Test -22 (SNOT-22) | Up to 7 months after treatment.
  At peak pollen season after treatment.
Change in allergen specific S- antibody levels. | 4-8 weeks after treatment, 9-12 months after treatment
  IgE, IgG, IgG4
Incidence of adverse events graded as mild-moderate-severe | From first injection to 30 days after last injection.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Olaf Cardell, Professor, Principal Investigator — Karolinska University Hospital
Locations (3):
- Sweden (3):
  - Allergy Unit, Södra Älvsborgs Hospital, Borås
  - ENT department, Skånes University Hospital Malmö and Lund, Malmo
  - ENT department, Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Senti G, Prinz Vavricka BM, Erdmann I, Diaz MI, Markus R, McCormack SJ, Simard JJ, Wuthrich B, Crameri R, Graf N, Johansen P, Kundig TM. Intralymphatic allergen administration renders specific immunotherapy faster and safer: a randomized controlled trial. Proc Natl Acad Sci U S A. 2008 Nov 18;105(46):17908-12. doi: 10.1073/pnas.0803725105. Epub 2008 Nov 10. PMID 19001265
- [Result] Hylander T, Latif L, Petersson-Westin U, Cardell LO. Intralymphatic allergen-specific immunotherapy: an effective and safe alternative treatment route for pollen-induced allergic rhinitis. J Allergy Clin Immunol. 2013 Feb;131(2):412-20. doi: 10.1016/j.jaci.2012.10.056. PMID 23374268
- [Result] Witten M, Malling HJ, Blom L, Poulsen BC, Poulsen LK. Is intralymphatic immunotherapy ready for clinical use in patients with grass pollen allergy? J Allergy Clin Immunol. 2013 Nov;132(5):1248-1252.e5. doi: 10.1016/j.jaci.2013.07.033. Epub 2013 Sep 13. No abstract available. PMID 24035151
- [Derived] Hellkvist L, Hjalmarsson E, Weinfeld D, Dahl A, Karlsson A, Westman M, Lundkvist K, Winqvist O, Georen SK, Westin U, Cardell LO. High-dose pollen intralymphatic immunotherapy: Two RDBPC trials question the benefit of dose increase. Allergy. 2022 Mar;77(3):883-896. doi: 10.1111/all.15042. Epub 2021 Aug 29. PMID 34379802